CLINICAL TRIAL: NCT04413461
Title: Efficiency of Trans-cutanéous Electrical Nerve Stimulation for Isolated Primary Enuresis : A Randomised Controlled Trial
Brief Title: Comparative Study of the Efficacy of TENS Versus Placebo in Isolated Primary Enuresis
Acronym: TENS-Enuresis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 19-HPNCL-03
Record Dates: First submitted 2020-05-22; First posted 2020-06-04 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Enuresis, Nocturnal
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TENS (Experimental)
  Interventions: Other: TENS
- TENS Sham (Placebo Comparator)
  Interventions: Other: TENS Sham

INTERVENTIONS:
Other: TENS — Transcutaneous Electro Neuro Stimulation
  Arms: TENS
Other: TENS Sham — placebo of Transcutaneous Electro Neuro Stimulation : similar device without electro stimulation
  Arms: TENS Sham

SUMMARY:
Nocturnal enuresis is a functional urinary disorder in children. It is intermittent urinary incontinence during sleep in children aged 5 years and older. It is said to be "primary" if the child has never been clean at night for at least 6 months and "isolated" if there are no other associated urinary symptoms, including daytime symptoms.

It is a common condition with significant repercussions, including disruption of family and social life and a frequent decline in self-esteem. Without treatment, it can persist into adulthood. All these reasons justify taking care of these children.

This is usually based on:

The establishment of hygienic-dietetic rules: Regular urination and before sleeping, limitation of fluid intake in the evening. They are systematically implemented, whatever the subsequent management Drug treatments (Desmopressin, oxybutynin). These treatments have an efficiency of 60 to 70% at 6 months post treatment and sometimes have side effects.

Non-drug treatments: Night-time "pee stop" alarms. They have an efficiency of around 70%. They are little used because they often wake up the whole family and are not reimbursed by social security.

TENS (Transcutaneous Electro Neuro Stimulation) is a neuro-modulation technique which consists of stimulating the nerves by means of skin electrodes in order to obtain a somatic response.

In urology, it is mainly used by stimulating either the sacral region, origin of the vesical innervation, or the tibial nerve. Its main indication is overactive bladder, a source of discomfort and incontinence.

It is used at home, the side effects are exceptional and it does not disturb the activities of the patients.

Few studies have evaluated its effectiveness in isolated primary enuresis.

DETAILED DESCRIPTION:
Nocturnal enuresis is a functional urinary disorder in children. It is intermittent urinary incontinence during sleep in children aged 5 years and older. It is said to be "primary" if the child has never been clean at night for at least 6 months and "isolated" if there are no other associated urinary symptoms, including daytime symptoms.

It is a common condition with significant repercussions, including disruption of family and social life and a frequent decline in self-esteem. Without treatment, it can persist into adulthood.

All these reasons justify taking care of these children.

This is usually based on:

The establishment of hygienic-dietetic rules: Regular urination and before sleeping, limitation of fluid intake in the evening. They are systematically implemented, whatever the subsequent management Drug treatments (Desmopressin, oxybutynin). These treatments have an efficiency of 60 to 70% at 6 months post treatment and sometimes have side effects.

Non-drug treatments: Night-time "pee stop" alarms. They have an efficiency of around 70%. They are little used because they often wake up the whole family and are not reimbursed by social security.

TENS (Transcutaneous Electro Neuro Stimulation) is a neuro-modulation technique which consists of stimulating the nerves by means of skin electrodes in order to obtain a somatic response.

In urology, it is mainly used by stimulating either the sacral region, origin of the vesical innervation, or the tibial nerve. Its main indication is overactive bladder, a source of discomfort and incontinence.

It is used at home, the side effects are exceptional and it does not disturb the activities of the patients.

Main objective is to compare the effectiveness of treatment with TENS versus TENS sham procedure (placebo) in isolated primary enuresis, one month after the end of treatment in patients from 5 to 17 years old The effectiveness will be evaluated by the evolution of the number of wet nights

ELIGIBILITY:
Inclusion Criteria:

Children 5 to 17 years old

* Medium or severe isolated primary enuresis (more than 1 episode per week)
* Never treated or in failure of previous treatment (with treatment discontinuation for at least 1 month)
* Affiliation to a social security scheme
* Good understanding of the protocol
* Signature of informed consent by a parent or the legal representative of parental authority

Exclusion Criteria:

Other pathologies which can influence urination behavior (Daytime urinary disorders)

* Treatment in progress which can modify voiding behavior
* TENS treatment in progress for another pathology

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
effectiveness of treatment with Transcutaneous Electro Neuro Stimulation (TENS) versus TENS sham procedure at 1 month post treatment | at 2 months
  The effectiveness will be evaluated by the evolution of the number of wet nights.
  Measure of number of wet nights per week at baseline before treatment by TENS and at 1 month after the end of treatment

SECONDARY OUTCOMES:
effectiveness of treatment with TENS versus TENS sham procedure at 1 month | at 1 month
  measure of number of wet nights per week at the end of treatment
quality of life during treatment | at baseline and at 1 month and at 2 month
  measure of quality of life with the Pediatric Quality of Life Inventory (Peds QL) questionnaire.
  The Pediatric Quality of Life Inventory (PedsQL) is a 23-items generic health status instrument with parent and child forms that assesses five domains of health (physical functioning, emotional functioning, psychosocial functioning, social functioning, and school functioning) in children and adolescents ages 2 to 18.
  For ease of interpretability, items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better HRQOL (Health-Related Quality of Life). The minimum value is 0 and maximum is 100.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CH de Cannes, Cannes
  - CH de GRASSE, Grasse
  - CHU de Nice, Nice
  - Hôpitaux Pédiatrique de Nice CHU Lenval, Nice

IPD SHARING:
Plan to Share IPD: No